CLINICAL TRIAL: NCT05024851
Title: Psychogenic and Neurogenic Components in Patients With Psychogenic or Neuropathic Pruritus : PRURINEURO, a Pilot Study
Brief Title: Psychogenic and Neurogenic Components in Patients With Psychogenic or Neuropathic Pruritus
Acronym: PRURINEURO
Status: Terminated | Type: Observational
Why Stopped: DECISION OF THE COORDINATOR
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PRURINEURO (29BRC21.0135)
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pruritus; Psychogenic Skin Disease; Neuropathic Pain; Itch
Keywords: Psychogenic Pruritus; Neuropathic Pruritus; Psychogenic Component; Neurogenic Component
MeSH Terms: conditions — Pruritus; Neuralgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Psychogenic pruritus
  Interventions: Other: Questionnaires
- Patients with Neuropathic Pruritus
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Evaluation of the Psychogenic and Neurogenic Components using questionnaires

SUMMARY:
Scientific research on pruritus is in intensive development, with significant advances in understanding its pathophysiology. The causes of pruritus are very huge; they can be classified into different categories; we can find dermatological causes, systemic causes, neuropathic or neurological causes, psychogenic or even idiopathic causes.

The diagnosis of psychogenic pruritus is often over stated, when no cause is found; therefore, it is important to see what is really relieving from psychic so as not to over-diagnose and adopt a therapy more in line with the real problem of the patient. In daily practice, it seems to have a tendency to separate psychogenic and neurogenic etiologies in the diagnosis of neuropathic or psychogenic pruritus.

In the case of patients with psychogenic pruritus and neuropathic pruritus, no study has attempted to study the respective part of psychogenic and neurogenic components. Consequently, it would therefore be interesting to assess the areas of superposition and distinction of neuropathic and psychogenic pruritus.

The aim of this pilot study is to assess the psychogenic and neurogenic components of psychogenic pruritus and neuropathic pruritus in order to improve understanding of the mechanism and therefore their management.

The main objective of this study is to highlight the differences and the potential common characteristics between psychogenic and neuropathic pruritus in order to improve the differential diagnosis between these two pathologies.

The secondary objective of this study is to describe the psychogenic and neurogenic characteristics of psychogenic and neuropathic pruritus.

DETAILED DESCRIPTION:
PruriNeuro : Non-interventional single-center prospective study organized and practiced on humans for the development of medical knowledge, in which the data are obtained by validated questionnaires.

The duration of participation is estimated at 1 hour.

Questionnaires used :

* Critères diagnostiques du prurit psychogène (Diagnosis criteria of functional itch disorder or psychogenic pruritus, from the French psychodermatology group)
* NP5 questionnaire
* Questionnaire de Brest
* HADS
* TAS-20
* DN4i

ELIGIBILITY:
Inclusion Criteria:

* Major (> 18 years old)
* Diagnosis of psychogenic pruritus or neuropathic pruritus made in consultation, in day hospital or in hospital, within the dermatology department at the CHRU de Brest
* Able to understand and agree to sign the information and non-opposition notice
* No opposition of the patient

Exclusion Criteria:

* Patient under legal protection (guardianship, curatorship)
* Minor (<18 years old)
* Acute or chronic condition which could limit the patient's ability to the study's participation
* Inability to understand and sign the information and non-opposition notice
* Refusal to give no opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuropathic or psychogenic pruritus consulting in the dermatology department of the CHRU de Brest.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Questionnaire de Brest | at the enrollment
  Qualitative assessment of pruritus, specifying the chronology, location, intensity, characteristics and effect on daily activities of the itching induced by pruritus
HADS (Hospital Anxiety and Depression Scale) | at the enrollment
  Total score for Depression or Anxiety 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
NP5 | at the enrollment
  A score of two criteria out of five is optimal to discriminate Neuropathic pruritus (NP) from Non-NP
TAS-20 | at the enrollment
  The TAS-20 is a self-report scale that is comprised of 20 items. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. There are 5 items that are negatively keyed (items 4, 5, 10, 18 and 19). The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
DN4i | at the enrollment
  score equal to or greater than 3 : in favor of neuropathic pruritus
Diagnosis criteria of functional itch disorder or psychogenic pruritus, from the French psychodermatology group | at the enrollment
  three compulsory criteria; Three additional criteria from seven items should also be present

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two years and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.